CLINICAL TRIAL: NCT00428155
Title: A Randomized Trial of Angioseal and Starclose for Hemostasis After PCI
Brief Title: Arterial Closure Device Comparison Trial II - ACDC Trial II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SMH#06-140
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-01-29 (Estimated); Status verified 2007-01

CONDITIONS: Arterial Hemostasis After Coronary Intervention
Keywords: hemostasis; angioplasty; stenting; closure device; angioseal; starclose

INTERVENTIONS:
Device: closure device placement

SUMMARY:
PCI (coronary angioplasty) is a procedure performed through a catheter to open up blockages in the coronary arteries using balloons and stents for the treatment of angina or myocardial infarction. The balloon catheters and stents are moved to the coronary arteries through a "sheath" (a small tube used for placing of balloon and stent catheters in the body) placed in a major artery passing through the groin. After the PCI procedure and the removal of sheath, an "arterial closure device" is commonly placed to stop bleeding and allow you to get out of bed sooner. Although the usefulness of "closure devices" has been documented before their approval by the regulatory authorities, it is unclear if one device is better compared to other commercially available devices.

The purpose of the study is to compare the two approved arterial closure devices, "Angioseal" and "Starclose". This study will help us identify the better of the two devices to improve patient comfort after the procedure.

DETAILED DESCRIPTION:
All patients scheduled to undergo percutaneous coronary interventions will be screened for inclusion into the study. Informed consent will be obtained and patients will be randomized to the placement of either Angioseal or a Starclose vascular closure device to achieve hemostasis after the PCI procedure. The randomization will take place after a femoral angiogram has confirmed the suitability of the femoral artery for placement of arterial closure device. All patients will be monitored for bleeding or hematoma formation for twelve hours after the procedure. Patients will be ambulated at two hours after placement of the arterial closure device. A complete blood count and a vascular ultrasound will be performed in all patients before discharge to assess blood loss and detect vascular complications such as hematoma, arteriovenous fistula or femoral artery pseudoaneurysm. A written quality of life survey will be completed before discharge and at four weeks. A nursing survey will be completed by the nursing staff to determine nurse-sensitive outcomes and nurse resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non emergent PCI procedures with a 6F arterial sheath.
* Femoral artery anatomy favorable for the placement of an arterial closure device.

Exclusion Criteria:

* Emergency PCI
* End stage renal disease
* Prior arterial closure device use within 90 days.
* Symptomatic peripheral vascular disease.
* Arterial puncture of the superficial femoral artery.
* Suspected double wall puncture (puncture of anterior & posterior wall of femoral artery).
* Placement of intra aortic balloon pump.
* Placement of a femoral venous sheath.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448
Dates: Start 2007-01

PRIMARY OUTCOMES:
A composite of major vascular complications defined as device failure, bleeding, large hematoma, local infection etc.

SECONDARY OUTCOMES:
Time to hemostasis
Lack of ambulation per protocol
Need for additional measures to achieve hemostasis (manual pressure, femostop use, etc.)
Minor vascular complication (minor bleeding, analgesic use)
post procedural myocardial infarction
30 day incidence of death, MI, TVR
Patient discomfort
Quality of life measurements at discharge and four weeks
Nurse resource utilization at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Asim Cheema, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada